CLINICAL TRIAL: NCT00484406
Title: Matrix Metalloproteinase Genetic Polymorphisms and Outcome of Non-ST Elevated Acute Coronary Syndromes
Brief Title: MMP Polymorphisms and Acute Coronary Syndromes
Status: Completed | Type: Observational
Sponsor: University of Trieste (Other)
Other Study IDs: FT-05-CG-201040106
Record Dates: First submitted 2007-06-07; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-05

CONDITIONS: Unstable Angina
Keywords: Matrix Metalloproteinases; Atherosclerosis; Genetic polymorphism; Acute coronary syndromes
MeSH Terms: conditions — Angina, Unstable; Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Some Matrix Metalloproteases, proteases degrading the extracellular matrix, play a relevant role in structure and stability of atherosclerotic plaques. Atherosclerotic plaques triggering acute coronary syndromes show increased expression of MMP-1, MMP-3 and MMP-9. Regulation of these MMPs is plaid by genetic polymorphisms, G+/G- at -1563 for MMP-1, 4A/5A- at -1612 for MMP-3, and a microsatellite (13-27 CA repeats around -90) for MMP-9.

It is conceivable that these polymorphisms correlate with the clinical outcome of acute coronary syndromes, particularly with those without ST segment Elevation (NSTEACS).

DETAILED DESCRIPTION:
Non-ST elevation acute coronary syndrome (NSTEACS) is a syndrome encompassing a spectrum of clinical manifestations between ischemic heart disease and acute myocardial infarction. It represents an important cause of morbidity and hospitalization in western countries: its incidence is estimated around 2/1000 subjects/year and about 10% of patients with acute coronary syndrome develop an acute myocardial infarction within 6 months. Another reason of concern is that patients require an invasive treatment, usually PTCA or CABG. ACS encompasses features of both an inflammatory and thrombotic disease; their abnormalities could be critical for evolution and complication of acute coronary syndrome.

Many inflammatory and coagulation indicators have been investigated, although the critical factors responsible for complications in NSTEACS remain elusive.

Matrix remodeling and consequent erosion or fissuration of the unstable plaque is supposed to be a key step of the development of acute coronary syndromes.

Neutral matrix metalloproteinases 1, 3 and 9 have been demonstrated to be actively produced in atherosclerotic tissue, compared to unaffected arteries. Mechanisms responsible for such increased expression might be related to inflammation, but also genetic regulation could account for an increased expression leading to a different clinical outcome of the syndrome.

Genetic polymorphisms are described for all three MMPs involved in ACS. MMP-1 insertion of a G in position creates an ets binding site that induces an eight times increase of the synthesis rate. For MMP-3 (stromelysin) polymorphism, a deletion of an A (adenosine) in position -1171 doubles the transcription activity and has been recently associated with acute myocardial infarction and progression of coronary stenosis. In MMP-9 a more complex polymorphism involves a microsatellite (AC) repeat in position -90 to -131. The mechanism leading to increased MMP-9 expression is probably related to the transition to Z-DNA within the microsatellite, which eases transcription. In vitro studies show that the longer the tandem repeats sequence, the higher the transcription.

No studies on metalloproteinase polymorphism in NSTEACS have been carried out, so far.

This study has been planned to assess if patients admitted to the hospital for NSTEACS could be associated to a different in hospital clinical outcome according to the genetic polymorphism of these proteases.

ELIGIBILITY:
Inclusion Criteria:

* non ST elevation acute coronary syndrome (NSTE ACS)

Exclusion Criteria:

* STE acute myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola FIOTTI, MD, Principal Investigator — University of Trieste, ITALY; Carlo Giansante, MD, Study Chair — University of Trieste, ITALY
Locations (2):
- Italy (2):
  - Azienda per i Servizi Sanitari n.6 "FRIULI OCCIDENTALE", Pordenone, Pordenone
  - Clinica Medica - University of Trieste, Trieste, Trieste

REFERENCES:
- [Background] Fiotti N, Altamura N, Fisicaro M, Carraro N, Uxa L, Grassi G, Torelli L, Gobbato R, Guarnieri G, Baxter BT, Giansante C. MMP-9 microsatellite polymorphism and susceptibility to carotid arteries atherosclerosis. Arterioscler Thromb Vasc Biol. 2006 Jun;26(6):1330-6. doi: 10.1161/01.ATV.0000219233.31702.c9. Epub 2006 Mar 30. PMID 16574900
- [Background] Galis ZS, Sukhova GK, Lark MW, Libby P. Increased expression of matrix metalloproteinases and matrix degrading activity in vulnerable regions of human atherosclerotic plaques. J Clin Invest. 1994 Dec;94(6):2493-503. doi: 10.1172/JCI117619. PMID 7989608
- [Background] Pollanen PJ, Lehtimaki T, Mikkelsson J, Ilveskoski E, Kunnas T, Perola M, Penttila A, Mattila KM, Nikkari ST, Syrjakoski K, Karhunen PJ. Matrix metalloproteinase3 and 9 gene promoter polymorphisms: joint action of two loci as a risk factor for coronary artery complicated plaques. Atherosclerosis. 2005 May;180(1):73-8. doi: 10.1016/j.atherosclerosis.2004.10.041. Epub 2004 Dec 18. PMID 15823277
- [Background] Terashima M, Akita H, Kanazawa K, Inoue N, Yamada S, Ito K, Matsuda Y, Takai E, Iwai C, Kurogane H, Yoshida Y, Yokoyama M. Stromelysin promoter 5A/6A polymorphism is associated with acute myocardial infarction. Circulation. 1999 Jun 1;99(21):2717-9. doi: 10.1161/01.cir.99.21.2717. PMID 10351963
- [Derived] Fiotti N, Moretti ME, Bussani R, Altamura N, Zamolo F, Gerloni R, Ukovich L, Ober E, Silvestri F, Grassi G, Adovasio R, Giansante C. Features of vulnerable plaques and clinical outcome of UA/NSTEMI: Relationship with matrix metalloproteinase functional polymorphisms. Atherosclerosis. 2011 Mar;215(1):153-9. doi: 10.1016/j.atherosclerosis.2010.12.010. Epub 2010 Dec 21. PMID 21232745